CLINICAL TRIAL: NCT06626295
Title: Exercise-snacks: an Effective Solution for Breaking the Sedentary Lifestyle and Improving the Physical Fitness of Obese Adolescents?
Brief Title: Exercise-snacks for Breaking the Sedentary Lifestyle and Improving the Physical Fitness of Obese Adolescents?
Acronym: SNACKEX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Avignon (Other)
Collaborators: Institut Saint Pierre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AU_ISP1_2024
Record Dates: First submitted 2024-09-23; First posted 2024-10-03 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Obese Adolescents; Sedentary Time; Exercise
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- exercise-snack group (Experimental): Exercise program:
  Adolescents in the exercise-snacks group will perform 4 "exercise-snacks" sessions per day during 3 weeks in addition to multidimensional care program. These sessions will consist of 1-min various intense supervised exercises . They will also receive information about their attitudes to physical activity.
  Interventions: Other: exercise-snack group
- control group (No Intervention): only the multidimensional care program without 'exercise-snacks'

INTERVENTIONS:
Other: exercise-snack group — Adolescents in the exercise-snacks group will perform 4 &#34;exercise-snacks&#34; sessions per day during 3 weeks in addition to multidimensional care program. These sessions will consist of 1-min various intense supervised exercises . They will also receive information about their attitudes to physical activity.
  Arms: exercise-snack group

SUMMARY:
The management of a person with obesity involves long-term behavioral changes with a balanced diet in both quantity and quality, along with the adoption of a more active lifestyle: increasing physical activities and reducing sedentary behaviors. The school setting has been identified as a favorable environment for interventions aimed at reducing and interrupting the time adolescents spend sitting and preventing the associated negative health consequences.

Recently, very short (< 1 minute) and intense exercises, called 'exercise-snacks,' have been reported to be effective in adults for 1) improving physical fitness over 6 weeks, and 2) improving vascular function and lowering blood glucose levels over a single day. Additionally, in adolescents with diabetes, they have been shown to reduce body fat. This raises the question of whether adding 'exercise-snack' sessions to a multidimensional care program for hospitalized obese adolescents could further improve their physical fitness in the short and medium term.

The objective of this project is to compare the effects of a traditional multidimensional care program with the addition of 'exercise-snacks' to the same care program without 'exercise-snacks' on the physical fitness, body composition, vascular function, and physical activity and sedentary behaviors of obese children in the short and medium term. Thirty-six obese adolescents will be included. The 'exercise-snack' group will perform six exercise sessions per day for three weeks in addition to the standard care. The control group will receive only the standard care. Assessments of physical fitness, body composition, vascular health, and questionnaires on physical activity, sedentary behavior, and cognitive restraint will be conducted at the beginning and end of the three-week program, as well as 1 and 3 months after the end of the program.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index Z-score corresponding to stage 2 obesity,
* no weight loss of more than 5% of total body weight in the past 3 months,
* parental consent
* minor's acceptance

Exclusion Criteria:

* Contraindication to physical activity
* current participation in a clinical trial

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-09-09 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Changes in aerobic fitness: predicted VO2max | at inclusion, at the end of the 3-weeks program and 1 and 3 month following the end of the program
  Measured by the Spartacus 15-15 field test, an intermittent maximal running field test with prediction of VO2max:
  For girls: VO2max = last stage * 153.4433 + BMI * 58.64534 + âge * -2.701522-921.2878 For boys: VO2max = last stage * 153.4433 + 320.1583 + BMI * 58.64534 + âge * -2.701522-921.2878

SECONDARY OUTCOMES:
Changes in fat mass | from inclusion to the end of the 3-weeks program and 1 and 3 month following the end of the program
  measured by medical body composition analyzer mBCA SECA, in kg
Changes in body mass index in kg/m² | at inclusion, at the end of the 3-weeks program and 1 and 3 month following the end of the program
change in carotid extra-media thickness | at inclusion, at the end of the 3-weeks program and 1 and 3 month following the end of the program
  measured by echocardiography (Mylab, Esaote, Italie) and off-line analyses by CAROLAB, in mm
Changes in carotid intima-thickness | at inclusion, at the end of the 3-weeks program and 1 and 3 month following the end of the program
  measured by echocardiography (Mylab, Esaote, Italie) and off-line analyses by CAROLAB, in mm
Change from baseline in carotid compliance (mm²/mmHg) | From inclusion to the end of the 3-weeks program and 1 and 3 month following the end of the program
  measured by echocardiography (Mylab, Esaote, Italie) according to the variations of systolic and diastolic arterial diameters and pulse pressure (measured on the left arm by an automated system Omron)
Changes in eating behaviours traits | at inclusion, at the end of the 3-weeks program and 1 and 3 month following the end of the program
  measured by the Three-Factor Eating Questionnaire to assess three factors: the cognitive restraint scale (6 items), the emotional eating scale (6 items), and the uncontrolled eating scale (9 items) with a 4-point response scale.
  For the TFEQ scores, means are computed for each subscale and are transformed to correspond to a 0-100 scale score Higher scores indicate higher levels of restrained eating, disinhibited eating, and predisposition to hunger.
Changes in psychometric properties of physical activity and sedentary | from inclusion to the end of the 3-weeks program and 1 and 3 month following the end of the program
  measured by a 31 items self-administered questionnaire CAPAS-Q to assess the psychometric properties of the Children and Adolescents Physical Activity (PA) and Sedentar (SB) by-Questionnaire (Fillon et al 2022) Responses are quoted from 1 to 4 for PA and from 1 to 6 for SB. The sum of items 1, 3, 6, 8, 10, 12, and 17 exploring PA duration, the sum of items 2, 4, 7, 11, 13, and 18 exploring PA intensity, within its different contexts of practice: school PA (i.e., the sum of items 1,2,3,4,5), non-school PA (the sum of items 6 to 14), and sports and leisure PA (the sum of items 15 to 18). The last 13 items designe to assess the SB dimension:, exploring screen ( the sum of items 2, 6, and 7) or non-screen non-screen ( the sum of items 1, 4, 5, 8, 9, 12 and 13) behaviors, the consecutive SB duration (the sum of items 3, 10 and 11) and the context of SB: school SB (the sum of items 1 to 3), non-school SB (the sum of items 4 to 11), SB during transportation (the sum of 12,13)
change in level of habitual physical activity | before inclusion and before the 1 and 3-month visit
  measured by accelerometric data using AX3, Axivity over 7-days consecutive period before inclusion and before the 1 and 3-month visit

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Instiutut Saint Pierre, Palavas-les-Flots
  - Institut Saint Pierre, Palavas-les-Flots

IPD SHARING:
Plan to Share IPD: No